CLINICAL TRIAL: NCT05642780
Title: A Multicenter, Open-label, Phase 2, Basket Study to Evaluate the Efficacy and Safety of SKB264 in Combination With Pembrolizumab in Subjects With Selected Solid Tumors
Brief Title: SKB264 in Combination With Pembrolizumab in Subjects With Selected Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Klus Pharma Inc. (Industry)
Collaborators: Myriad Genetics, Inc. (Industry); Discovery Life Sciences, LLC (Unknown); Ventana Medical Systems, Inc (Unknown); Frontage Laboratories, Inc. (Unknown); Clario (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-II-06
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- cohort A (Experimental): subjects will receive SKB264 in combination with pembrolizumab by intravenous administration
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- cohort B (Experimental): subjects will receive SKB264 in combination with pembrolizumab by intravenous administration
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- cohort C (Experimental): subjects will receive SKB264 in combination with pembrolizumab by intravenous administration
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- cohort D (Experimental): subjects will receive SKB264 in combination with pembrolizumab by intravenous administration
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- Cohort E (Experimental): subjects will receive SKB264 in combination with pembrolizumab by intravenous administration
  Interventions: Drug: SKB264; Drug: Pembrolizumab

INTERVENTIONS:
Drug: SKB264 — be administrated as an intravenous (IV) infusion on Day 1,15, 29 of each 42-day cycle;
Drug: Pembrolizumab — be administrated as an intravenous (IV) infusion on Day 1 of each 42-day cycle;
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combination of SKB264 and Pembrolizumab in patients with selected solid tumors including cervical cancer, urothelial cancer, ovarian cancer, prostate cancer,advanced endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 .
2. Subjects with expected survival ≥ 3 months.
3. Cohort A: Subjects with recurrent or metastatic cervical cancer
4. Cohort B: Subjects with locally advanced or metastatic urothelial carcinoma
5. Cohort C: Subjects with recurrent ovarian cancer
6. Cohort D: Subjects with metastatic prostate cancer
7. Subjects have at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
8. Subjects able to provide tumor blocks or slides for biomarker test.
9. Subjects have relatively good organ function and bone marrow function.
10. Subjects must have recovered from all toxicities from previous therapy with the exception of toxicities not considered a safety risk.
11. Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
12. Subject is capable of giving signed informed consent.
13. Cohort E: Subjects with advanced endometrial cancer.

Exclusion Criteria:

1. Subjects with active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis are not eligible.
2. Subjects who suffer from cardiovascular diseases of clinical significance.
3. Subjects with serious and/or uncontrolled concomitant diseases.
4. Subjects diagnosed active hepatitis B or hepatitis C.
5. Subjects have known human immunodeficiency virus (HIV) infection that is not well controlled.
6. Subjects with known active tuberculosis.
7. Known allergy or hypersensitivity to pembrolizumab or SKB264, or the excipients of pembrolizumab or SKB264.
8. Subjects with history of allogeneic tissue/solid organ transplant.
9. Subjects previously treated with TROP2 targeted therapy.
10. Subjects who are vaccinated with live vaccine within 30 days before the first dose, or plan to be vaccinated with live vaccine during the study period.
11. Subjects participating in another clinical study, unless it is an observational (non-intervention) clinical study or the follow-up period of an intervention study.
12. The Investigator considers other situations that will interfere with the evaluation of the study intervention or the safety of the subjects or the interpretation of the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and adverse events (AEs) | From subject sign the ICF to 30 days after the last dose of study treatment
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Objective Response Rate (ORR) | From baseline until disease progression, death or other protocol defined reason up to approximately 21 months
  ORR is defined as the proportion of subjects with confirmed CR or PR as the best overall response assessed per RECIST 1.1.
Prostate-specific antigen (PSA) response rate (Cohort D) | From baseline until disease progression, death or other protocol defined reason up to approximately 21 months
  The percentage of subjects in the analysis population who have a negative change (decrease) in PSA level of ≥ 50% measured twice ≥ 3 weeks apart

CONTACTS AND LOCATIONS:
Locations (48):
- United States (8):
  - Community Clinical Research Center, Anderson, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Anne Arundel Medical Center (AAMC), Annapolis, Maryland
  - UT Health East Texas - Hope Cancer Center Tyler, Tyler, Minnesota
  - Westchester Medical Center, Hawthorne, New York
  - Texas Oncology, P.A. Amarillo, TX, Amarillo, Texas
  - Texas Oncology, P.A. Austin, TX, Austin, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc. Roanoke, VA, Roanoke, Virginia
- Australia (3):
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Flinders Medical Centre, Bedford Park
  - Wollongong Hospital, Kogarah
- Belgium (3):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (2):
  - BC Cancer - Kelowna, Kelowna, British Columbia
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal
- China (29):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jinlin
  - The Second Hospital of Dalian, Dalian, Liaoning
  - Weifang People's Hospital, Weifang, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Qilu Hosptial of Qlilu University, Jinan
  - Shandong Cancer Hospital, Jinan
  - Nanjing Drum Tower Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Obstetrics and Gynecology Hospital Affiliated to Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Henan Cancer Hospital, Affiliated Cancer Hospital of Zhengzhou Universit, Zhengzhou
  - Henan Cancer Hospital, Zhengzhou
  - The first Affiliated Hospital of Zhengzhou University, Zhengzhou
- Poland (3):
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Pratia MCM Krakow, Krakow
  - Biokinetica S.A., Przychodnia Jozefow, Warsaw